CLINICAL TRIAL: NCT04226092
Title: Pre-SunBeam Pilot Study: Comparative Assessment of TEWL Measurements From AquaFlux vs. Handheld GPSkin Pro in Young Children With and Without AD
Brief Title: Pre-SunBeam TEWL AUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Jewish Health (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AP09162019
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Atopic Dermatitis
Keywords: Transepidermal Water Loss
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with atopic dermatitis (Experimental)
  Interventions: Device: GPSkin Barrier Pro; Device: Aquaflux AF200
- Control subjects (Experimental)
  Interventions: Device: GPSkin Barrier Pro; Device: Aquaflux AF200

INTERVENTIONS:
Device: GPSkin Barrier Pro — This study is a pilot study to determine if this device produces similar readings than Aquaflux AF200 for TEWL/skin barrier on patients with and without atopic dematitis (AD).
Device: Aquaflux AF200 — This study is a pilot study to determine if this device produces similar readings than GPSkin Barrier Pro for TEWL/skin barrier on patients with and without atopic dematitis (AD).

SUMMARY:
Transepidermal Water Loss (TEWL) measurements are a valuable tool to determine the integrity of a person's skin barrier. In patients with skin conditions, like atopic dermatitis, skin barrier can be disrupted or weakened, leading to a more severe phenotype and disease characteristics. There are several commercially available TEWL measuring devices, including the Aquaflux AF200 and the GPSkin Barrier Pro. This study is a pilot study to determine if these two devices produce similar readings for TEWL/skin barrier on patients with and without atopic dematitis (AD). The research team would like to investigate whether these devices are comparable for initial TEWL readings as well as after several rounds of tape strips have been collected from the skin. Tape strips are small circular adhesives, much like tape, that remove the very outermost layers of skin cells. It will be important to know if both of these devices provide correlative values for TEWL once the outermost layers of the skin have been removed by tape stripping.

ELIGIBILITY:
Inclusion Criteria:

1. Parent guardian must be able to understand and provide informed consent and participant provide assent as applicable per Institutional Review Board (IRB) guidelines and regulations.
2. Male or female, less than or equal to 3 years of age inclusive at Screening
3. Active AD using Standard Diagnostic Criteria (AAD criteria, Eichenfield et al, 2014). Participant must have an area of non-lesional AD (EASI of 0) within 5 cm. of the measured lesional area within the same region. Participant must have lesional and nonlesional areas of at least 3 cm in diameter to allow for both devices to be tested in contiguous areas OR FOR HEALTHY CONTROLS
4. Participant must meet all of the following criteria:

   1. No personal history or current manifestations of AD; no current food allergy, asthma, allergic rhinitis (based on self-report)
   2. No evidence of dry skin or other skin issue (EASI score of 0)

Exclusion Criteria:

1. Inability or unwillingness of a parent guardian to give written informed consent, or participant to give assent, if applicable, or to comply with study protocol
2. Who have any skin disease other than AD that might compromise the stratum corneum barrier in infants and young children (e.g., ichthyosis, psoriasis, extensive seborrheic dermatitis, scabies)
3. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
4. Use of any topical product (e.g., emollient, topical corticosteroids, topical immunomodulatory agents, topical antibiotics) on extremity for testing within 2 hours of the Enrollment Visit.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of TEWL curves | baseline
  Correlation in TEWL curve (AUC) between two TEWL devices (Aquaflux AF200 and GPSkin Barrier Pro) in non-lesional atopic dermatitis and healthy skin.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Northwestern University/Lurie Children's Hosptial, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No